CLINICAL TRIAL: NCT02240147
Title: Start-to-Sport - Feasibility and Efficacy of Individualized, Telemonitored, Home-based Exercise for Adolescents and Adults With Congenital Heart Disease
Brief Title: Start-to-Sport - Home-based Exercise for Adolescents and Adults With Congenital Heart Disease
Acronym: S2S-ACHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Roselien Buys, Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2S-ACHD
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Congenital Heart Defect
Keywords: adult congenital heart disease; exercise capacity; exercise training; physical activity
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- home-based exercise training (Experimental)
  Interventions: Behavioral: home-based exercise training
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: home-based exercise training — During a 30 minute face-to-face motivational interview with an exercise specialist, the patient will be advised and coached about his exercise prescription, on how to implement it in his own daily life and on how to prevent relapse. Furthermore, the patients will receive instructions on how to monitor their exercise intensity and on recognizing adverse signals. During the following 12 weeks, patients will be asked to exercise 4.5 hours per week within the prescribed exercise intensity range according to the guidelines.
  Arms: home-based exercise training

SUMMARY:
Almost 1% of all baby's is born with a heart defect (CHD) and most of them survive. Even though outcomes are good, they need lifelong follow-up because of a higher risk for cardiovascular diseases. Studies have shown that patients with CHD are not active enough and that a substantial amount of patients is overweight. Hence preventive strategies and education should not only focus on the heart problem, but also on a healthy lifestyle including physical activity. Recently a new guideline introduced exercise prescription based on the absence/presence of certain key elements. However, a number of important questions remain that preclude implementation in clinical practice. Therefore a 'Start-to-Sport' program for adults with CHD, based on this new guideline, will be investigated. This study is a randomized controlled trial that investigates the effects of the program on daily physical activity, exercise capacity, quality of life and exercise self-efficacy both in short (12 weeks) and long (52 weeks) term, along with possible mechanisms for the training effects by using a new exercise-testing protocol that looks simultaneously to all body parts that are involved during exercise. Ultimately, our findings will result in the implementation of the guideline in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* adolescents and adults with congenital heart disease
* 16 to 65 years

Exclusion Criteria:

* congenital rhythm or conduction disorders
* isolated congenital coronary artery anomalies
* pregnancy
* being listed for heart transplantation
* inability to perform standard physical activities due to mental/physical disability.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
peak oxygen uptake | baseline, post-intervention, after 1 year

SECONDARY OUTCOMES:
physical activity | baseline, post-intervention and after 1 year
  Physical activity will be assessed by means of the Sensewear mini armband. The patient will be asked to wear the device day and night during 1 week, while also taking notes of the physical activities undertaken by means of a logbook.

CONTACTS AND LOCATIONS:
Overall Officials: Roselien Buys, PhD, Principal Investigator — KU Leuven; Werner Budts, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Budts W, Borjesson M, Chessa M, van Buuren F, Trigo Trindade P, Corrado D, Heidbuchel H, Webb G, Holm J, Papadakis M. Physical activity in adolescents and adults with congenital heart defects: individualized exercise prescription. Eur Heart J. 2013 Dec;34(47):3669-74. doi: 10.1093/eurheartj/eht433. Epub 2013 Nov 7. No abstract available. PMID 24204010